CLINICAL TRIAL: NCT01266629
Title: The Clinical Utility of Fecal Calprotectin and Lactoferrin in Patients Undergoing Capsular Endoscopy: A Prospective Study
Brief Title: The Clinical Utility of Fecal Caprotectin and Lactoferrin in Patients Undergoing Capsular Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Ariella Shitrit Shaare Zedek Medical Center, Shaare Zedek Medical Center
Other Study IDs: 2010-147
Record Dates: First submitted 2010-12-23; First posted 2010-12-24 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-10

CONDITIONS: Crohn's Disease
Keywords: small bowel
MeSH Terms: conditions — Crohn Disease

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- capsule patients: All patients that will undergo endoscopic capsule

SUMMARY:
Capsule endoscopy (CE) is considered as a gold standard examination for small bowel Crohn's disease. However, it is time-consuming, expensive and results are largely influenced by the operator's skills. We, therefore, want to assess the predictive value of fecal calprotectin and lactoferrin in patients undergoing CE.

DETAILED DESCRIPTION:
Capsule endoscopy (CE), a novel and wireless method of investigating the small bowel uses a remote instrument that is swallowed and propelled through the gastrointestinal tract by the action of peristalsis. The capsule contains an imaging device, which transmits images of the intestine to sensors on the abdominal wall. It has the ability to detect diffuse mucosal disease but without the inadvertent radiation exposure. Numerous studies have compared the utility of small bowel radiology to CE for the investigation of Crohn's disease. A recent meta-analysis showed that CE is superior to small bowel radiology, CT enterography and ileo-colonoscopy in the setting of suspected Crohn's disease. Capsule endoscopy has now developed an established role in the investigation pathway of small bowel Crohn's disease. However CE requires placement of an eight-lead sensor array over the abdomen that receives image and localization data transmitted from the capsule. The current process of applying this array to the skin has several disadvantages: firstly, it is time-consuming; secondly, it can be cumbersome for the patient; and thirdly, it is often difficult to place the leads consistently. Moreover, CE is expensive and results are largely influenced by the operator's skills.

Among the available fecal biomarkers for the diagnosis and monitoring of inflammatory bowel disease (IBD), only calprotectin and lactoferrin have translated into useful clinical tools.

Calprotectin (MRP8/14) is a calcium-binding heterodimer of the S100 protein family, presents in granulocytes, macrophages, and epithelial cells of humans and other mammals.It is believed to play an essential role in immunity. Calprotectin is released upon neutrophil/monocyte activation, when it can be detected in serum and body fluids, including stool. It is poorly degraded during passage through the gastrointestinal tract and remains stable in refrigerated storage. Together, these features make calprotectin a potentially useful marker of clinical inflammatory and neoplastic states. Recently, several studies suggested that a high fecal calprotectin concentration may distinguish patients with inflammatory bowel disease (IBD) from patients with irritable bowel syndrome (IBS).

Lactoferrin (LF) is an iron binding glycoprotein secreted by most mucosal membranes and a major component of secondary granules of polymorphonuclear neutrophils, a component of the inflammatory response. A number of studies have investigated the use of lactoferrin as a non invasive marker in the distinction of inflammatory bowel disease (IBD) and non inflammatory conditions. Whilst a high sensitivity of LF has been reported for active IBD in comparison to IBS, the distinction of inactive IBD and IBS is less clear . Lactoferrin can be detected using simple and cheap techniques and it has excellent stability in feces over a long period of time. Fecal lactoferrin has a good diagnostic precision for separating organic and functional intestinal disease.

The aim of this prospective study is to assess the clinical utility of fecal calprotectin and lctoferrin in patients undergoing CE.

Exclusion criteria Intake of nonsteroidal agents and/or antibiotics during the three months preceding the study, concomitant serious illness, pregnancy, alcohol abuse, and evidence of a respiratory tract infection.

Study protocol After obtaining informed consent from the patients, data will collect on patient symptoms including the presence of abdominal pain, weight loss, diarrhoea, abdominal mass, extra-intestinal manifestations or family history of IBD. All patients will undergo a non diagnostic colonoscopy and gastro copy prior to CE referral.

Study protocol include diagnostic CE and stool examinations. Stool Analysis Prior to CE preparation, patients will ask to supply a stool specimen which they were to store in a household freezer and bring with them on the day of examination. The specimens will freeze at -20°C until assay. Fecal calprotectin levels will determine with a commercially available quantitative enzyme-linked immunoassay (Calpreset; Eurospital, Trieste, Italy and IBD SCAN) . Faecal lactoferrin test will perform on each thawed sample as previously described .Normal levels of calprotectin will define as 25 mg/kg stool.

Capsule endoscopy The description of CE is well reported in the literature (Pillcam SB, Given Imaging, Yoqneum,Ltd) .Patients will fast overnight for 12 hours after ingestion of two sachets of polyethylene glycol solution (Kleen-Prep, Norgine). Patients were allowed to drink 2 hours after and eat a light snack 4 hours after ingestion of the capsule.

Blood markers In addition, blood will collect from all patients for measurement of complete blood count, C-reactive protein (CRP) level, and erythrocyte sedimentation rate (ESR) by standard methods (normal values ESR <12 mm/h; CRP <5 mg/l).

Calprotectin and lactoferrin levels in stool will compare to the clinical and laboratory parameters.

ELIGIBILITY:
Inclusion Criteria:All consecutive patients referred for endoscopic capsule -

Exclusion Criteria:Intake of nonsteroidal agents and/or antibiotics during the three months preceding the study, concomitant serious illness, pregnancy, alcohol abuse, and evidence of a respiratory tract infection.

-

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients referred for capsule on an outpatient basis will include in the study. Indications for EC will be suspicion of crohn's disease, unexplained anemia, and bleeding, and abnormal findings in commuted tomography. All patients underwent non diagnostic colonoscopy and gastroscopy prior to EC referral.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2010-12; Primary Completion 2011-06 (Estimated); Study Completion 2011-09 (Estimated)

PRIMARY OUTCOMES:
correlations between capsule and fecal markers | end of the study
  To assess the correlations between positive fecal markers and abnormal findings in endoscopic capsule

SECONDARY OUTCOMES:
correlations between serum markers and capsule | end of the study
  correlations between CRP, ESR , PLT and abnormal findings in capsule

CONTACTS AND LOCATIONS:
Overall Officials: Ariella Shitrit, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (1):
- Shaare Zedek, Jerusalem, Israel

REFERENCES:
- [Derived] Bar-Gil Shitrit A, Koslowsky B, Livovsky DM, Shitrit D, Paz K, Adar T, Adler SN, Goldin E. A prospective study of fecal calprotectin and lactoferrin as predictors of small bowel Crohn's disease in patients undergoing capsule endoscopy. Scand J Gastroenterol. 2017 Mar;52(3):328-333. doi: 10.1080/00365521.2016.1253769. Epub 2016 Nov 13. PMID 27841040